CLINICAL TRIAL: NCT00544115
Title: A Phase II Trial of Allogeneic Peripheral Blood Stem Cell Transplantation From Matched Unrelated Donors in Patients With Advanced Hematologic Malignancies and Hematological Disorders
Brief Title: Donor Peripheral Stem Cell Transplant in Treating Patients With Advanced Hematologic Cancer or Other Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01089; P30CA033572 (NIH); CHNMC-01089; 01089; CDR0000566376 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Precancerous/Nonmalignant Condition
Keywords: graft versus host disease; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; atypical chronic myeloid leukemia; chronic myelomonocytic leukemia; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; secondary acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; childhood nasal type extranodal NK/T-cell lymphoma; recurrent childhood large cell lymphoma; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; recurrent childhood lymphoblastic lymphoma; Burkitt lymphoma; recurrent childhood small noncleaved cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; refractory chronic lymphocytic leukemia; refractory multiple myeloma; stage III multiple myeloma; aplastic anemia; paroxysmal nocturnal hemoglobinuria; adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage II multiple myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precancerous Conditions; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Extranodal NK-T-Cell; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Recurrence; Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Busulfan; Cyclophosphamide; Cyclosporine; Etoposide; fludarabine phosphate; Melphalan; Methotrexate; Mycophenolic Acid; Sirolimus; Tacrolimus; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

ARMS (6):
- Regimen I (Active Comparator): Patients undergo total body irradiation (TBI) on days -7 to -4 and receive cyclophosphamide IV on days -3 and -2. Alternatively, patients may receive cyclophosphamide on days -7 and -6 and undergo TBI on days -4 to -1.
  Interventions: Drug: cyclophosphamide; Drug: cyclosporine; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation
- Regimen II (Active Comparator): Patients receive busulfan IV over 2 hours once on day -8 and then every 6 hours on days -7 to -4. Patients also receive cyclophosphamide IV on days -3 and -2.
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Drug: cyclosporine; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation
- Regimen III (Active Comparator): Patients undergo TBI on days -7 to -4 and receive etoposide IV on day -3.
  Interventions: Drug: cyclosporine; Drug: etoposide; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation
- Regimen IV (Active Comparator): Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3 and melphalan IV on day -2.
  Interventions: Drug: cyclosporine; Drug: fludarabine phosphate; Drug: melphalan; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation
- Regimen V (Active Comparator): Patients receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo TBI on day 0.
  Interventions: Drug: cyclosporine; Drug: fludarabine phosphate; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation
- Regimen VI (Active Comparator): Patients receive busulfan IV over 3 hours and fludarabine phosphate IV over 30 minutes on days -5 to -2.
  Interventions: Drug: busulfan; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: methotrexate; Drug: mycophenolate mofetil; Drug: sirolimus; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: busulfan
  Arms: Regimen II; Regimen VI
Drug: cyclophosphamide
  Arms: Regimen I; Regimen II
Drug: cyclosporine
Drug: etoposide
  Arms: Regimen III
Drug: fludarabine phosphate
  Arms: Regimen IV; Regimen V; Regimen VI
Drug: melphalan
  Arms: Regimen IV
Drug: methotrexate
Drug: mycophenolate mofetil
Drug: sirolimus
Drug: tacrolimus
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: total-body irradiation
  Arms: Regimen I; Regimen III; Regimen V

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation before a donor peripheral stem cell transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving tacrolimus, methotrexate, cyclosporine, mycophenolate mofetil, and sirolimus before and after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well donor peripheral stem cell transplant works in treating patients with advanced hematologic cancer or other disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate hematopoietic recovery, using neutrophil and platelet engraftment as the primary criterion, in patients with advanced hematologic malignancies or other disorders undergoing allogeneic peripheral blood stem cell (PBSC) transplantation from matched unrelated donors.
* To evaluate the incidence of acute and chronic graft-versus-host-disease (GVHD) in patients undergoing allogeneic PBSC transplantation from matched unrelated donors.

Secondary

* To evaluate the impact of HLA class I and class II allele-matching on the incidence of GVHD and on the survival outcome of these patients.
* To evaluate overall survival, disease-free survival, and relapse in these patients.

OUTLINE: Patients are stratified according to type of conditioning regimen (myeloablative vs reduced-intensity myeloablative). Patients are assigned to a conditioning regimen according to diagnosis, age, disease status, prior radiotherapy, and prior autologous stem cell transplantation.

* Conditioning regimen:

  * Regimen I: Patients undergo total body irradiation (TBI) on days -7 to -4 and receive cyclophosphamide IV on days -3 and -2. Alternatively, patients may receive cyclophosphamide on days -7 and -6 and undergo TBI on days -4 to -1.
  * Regimen II: Patients receive busulfan IV over 2 hours once on day -8 and then every 6 hours on days -7 to -4. Patients also receive cyclophosphamide IV on days -3 and -2.
  * Regimen III: Patients undergo TBI on days -7 to -4 and receive etoposide IV on day -3.
  * Regimen IV: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3 and melphalan IV on day -2.
  * Regimen V: Patients receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo TBI on day 0.
  * Regimen VI: Patients receive busulfan IV over 3 hours and fludarabine phosphate IV over 30 minutes on days -5 to -2.
* Allogeneic peripheral blood stem cell (PBSC) transplantation: All patients undergo allogeneic PBSC transplantation on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive one of the following GVHD prophylaxis regimens:

  * Regimen A: Patients receive tacrolimus IV or orally on days -1 to 180 and methotrexate IV on days 1, 3, 6, and 11.
  * Regimen B: Patients receive cyclosporine IV or orally twice daily on days -1 to 180, mycophenolate mofetil IV over 2 hours or orally twice daily on days 0-27, and methotrexate IV on days 1, 3, and 6.
  * Regimen C: Patients receive tacrolimus IV continuously or orally, and oral sirolimus beginning on day -3. Patients also receive methotrexate IV on days 1, 3, and 6.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Acute lymphocytic leukemia (ALL), meeting one of the following criteria:

    * In first relapse or beyond
    * High-risk ALL, defined by any of the following:

      * Hypoploidy (≤ 44 chromosomes)
      * Pseudodiploidy with translocations or molecular evidence of t(9;22), 11q23, or t(8;14), excluding B-cell ALL
      * Elevated WBC at presentation (WBC > 20,000/mm³ [for patients > 18 years of age]; WBC > 200,000/mm³ [for patients 12-18 years of age])
  * Acute myeloid leukemia (AML), meeting one of the following criteria:

    * In first complete remission
    * Failed to achieve remission
    * In first relapse or beyond
    * Secondary AML (> 30% blasts in marrow aspirate)

      * Should receive induction chemotherapy to obtain remission, if possible, before transplant
  * Chronic myelogenous leukemia, meeting one of the following criteria:

    * In first or second chronic phase or accelerated phase
    * In blast crisis, defined as > 30% promyelocytes plus blasts in the bone marrow
  * Myelodysplastic syndromes, including any of the following:

    * Refractory anemia with excess blasts (RAEB)
    * Chronic myelomonocytic leukemia
    * RAEB in transformation
  * Refractory non-Hodgkin lymphoma, chronic lymphocytic leukemia, Hodgkin lymphoma, or multiple myeloma

    * Received and failed front-line therapy, high-dose therapy and autologous stem cell transplantation, or salvage therapy
  * Myeloproliferative disorders/myelofibrosis may be allowed on a case by case basis
  * Severe aplastic anemia, paroxysmal nocturnal hemoglobinuria, or any other hematologic disorder requiring transplantation
* Patients > 55 years of age with hematologic diseases treatable by allogeneic stem cell transplantation who are not eligible for IRB 99190 are eligible
* No uncontrolled CNS involvement of disease
* No matched (6/6) related donor available
* HLA-identical unrelated donor available

  * HLA-phenotypically identical for HLA-A and HLA-B alleles and identical for DRB1 alleles by DNA typing for both class I and class II antigens

    * Allele mismatch for HLA class I (i.e., B 2701 vs B 2702) allowed if no alternative donors
    * Allele mismatch for class II (i.e., DRB1 0401 vs 0402) or minor mismatch for class I cross reactive group (CREG) (i.e., A 2 vs A 28) allowed in patients ≤ 35 years of age requiring urgent transplant

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* Life expectancy > 8 weeks
* LVEF ≥ 45% at rest
* AST ≤ 2 times normal (unless liver function abnormality is due to underlying disease)
* Total bilirubin < 1.5 times normal (unless liver function abnormality is due to underlying disease)
* Creatinine ≤ 1.5 times normal OR creatinine clearance ≥ 60 mL/min
* DLCO ≥ 40% of predicted (corrected for hemoglobin)
* No coexisting medical problem that would significantly increase the risk of the transplant procedure
* HIV negative
* Not pregnant

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2001-10-16 (Actual); Primary Completion 2007-03-13 (Actual); Study Completion 2026-04-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Auayporn P. Nademanee, MD, Study Chair — City of Hope Comprehensive Cancer Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Among the 260 enrolled patients, who consented to the study, 5 patients were not eligible.
Groups:
- Regimen I: Patients undergo total body irradiation (TBI) on days -7 to -4 and receive cyclophosphamide IV on days -3 and -2. Alternatively, patients may receive cyclophosphamide on days -7 and -6 and undergo TBI on days -4 to -1.
  cyclophosphamide
  cyclosporine
  methotrexate
  mycophenolate mofetil
  sirolimus
  tacrolimus
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
- Regimen II: Patients receive busulfan IV over 2 hours once on day -8 and then every 6 hours on days -7 to -4. Patients also receive cyclophosphamide IV on days -3 and -2.
  busulfan
  cyclophosphamide
  cyclosporine
  methotrexate
  mycophenolate mofetil
  sirolimus
  tacrolimus
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
- Regimen III: Patients undergo TBI on days -7 to -4 and receive etoposide IV on day -3.
  cyclosporine
  etoposide
  methotrexate
  mycophenolate mofetil
  sirolimus
  tacrolimus
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
- Regimen IV: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -3 and melphalan IV on day -2.
  cyclosporine
  fludarabine phosphate
  melphalan
  methotrexate
  mycophenolate mofetil
  sirolimus
  tacrolimus
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
- Regimen V: Patients receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo TBI on day 0.
  cyclosporine
  fludarabine phosphate
  methotrexate
  mycophenolate mofetil
  sirolimus
  tacrolimus
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
- Regimen VI: Patients receive busulfan IV over 3 hours and fludarabine phosphate IV over 30 minutes on days -5 to -2.
  busulfan
  cyclosporine
  fludarabine phosphate
  methotrexate
  mycophenolate mofetil
  sirolimus
  tacrolimus
  allogeneic hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
Period: Overall Study
Arm/Group | Regimen I | Regimen II | Regimen III | Regimen IV | Regimen V | Regimen VI
Started | 62 | 17 | 130 | 4 | 40 | 2
Completed | 62 | 17 | 130 | 4 | 40 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen I | Regimen II | Regimen III | Regimen IV | Regimen V | Regimen VI | Total
Number analyzed (Participants) | 62 | 17 | 130 | 4 | 40 | 2 | 255
Age, Continuous [Median (Full Range); unit: years] | 38 [14 to 62] | 52 [12 to 62] | 50 [6 to 67] | 22 [18 to 42] | 37 [7 to 58] | 44 [41 to 47] | 44 [6 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 11 | 65 | 2 | 17 | 1 | 120
  Male | 38 | 6 | 65 | 2 | 23 | 1 | 135
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 0 | 8 | 1 | 2 | 0 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 3 | 1 | 0 | 0 | 4
  White | 55 | 17 | 118 | 2 | 38 | 2 | 232
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 1 | 0 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 62 | 17 | 130 | 4 | 40 | 2 | 255

OUTCOME MEASURES:

1. Primary Outcome: Neutrophil Engraftment - The Days Till ANC Recovery
Description: The primary engraftment endpoint, neutrophil engraftment, is defined as the first of three consecutive days on which the absolute neutrophil count is > 500/µL. The duration and extent of neutrophil engraftment is the time from transplant to neutrophil engraftment.
Time Frame: Up to 180 days post transplant
Population: Some patients had engraftment failure and some had missing data. Therefore, the overall number of participants analyzed in each regimen is less than the overall number in the Participant Flow module.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Regimen I | Regimen II | Regimen III | Regimen IV | Regimen V | Regimen VI
Number analyzed (Participants) | 42 | 13 | 113 | 3 | 36 | 1
days | 17 [11 to 39] | 16 [13 to 21] | 15 [8 to 36] | 14 [14 to 17] | 18 [11 to 28] | 16 [16 to 16]

2. Secondary Outcome: Two-year Overall Survival
Description: Overall survival (OS) was measured from peripheral stem cell infusion to death from any cause. It was estimated using the Kaplan-Meier method; the 95% confidence interval was calculated using Greenwood's formula. Participants were followed up to 2 years after transplant and Kaplan-Meier survival analysis was used to generate the two-year Overall Survival estimate presented.
Time Frame: Up to 2 years post transplant
Population: 1 subject in Regimen II did not have transplant.
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | Regimen I | Regimen II | Regimen III | Regimen IV | Regimen V | Regimen VI
Number analyzed (Participants) | 62 | 16 | 130 | 4 | 40 | 2
percentage of survival probability | 58 [45 to 69] | 50 [25 to 71] | 54 [45 to 62] | 50 [6 to 84] | 38 [23 to 52] | 50 [0.1 to 91]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to Day 100 post-transplant. All-Cause Mortality was assessed from start of protocol treatment to death due to any cause, or last follow-up, whichever comes first, assessed up to 20 years.
Arm/Group | Regimen I | Regimen II | Regimen III | Regimen IV | Regimen V | Regimen VI
All-Cause Mortality (participants affected / at risk) | 45/62 | 14/17 | 103/130 | 2/4 | 32/40 | 1/2
Serious Adverse Events (participants affected / at risk) | 4/62 | 1/17 | 7/130 | 0/4 | 3/40 | 1/2
Other Adverse Events (participants affected / at risk) | 14/62 | 4/17 | 38/130 | 0/4 | 10/40 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen I (N=62) | Regimen II (N=17) | Regimen III (N=130) | Regimen IV (N=4) | Regimen V (N=40) | Regimen VI (N=2)
Coagulation - Other (Specify, __) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage/bleeding associated with surgery, intra-operative or postoperative (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melena/GI bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein flow (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy for BMT studies, if specified by the protocol. (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea associated with GVHD for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, __) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight gain - Veno-Occlusive Disease (VOD) for BMT studies if specified in the protocol. (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilirubin associated with GVHD for BMT studies, if specified in the protocol. (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (Specify, __) (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Infection, Bacterial (COH) (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infection, Viral (COH) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkalosis (metabolic or respiratory) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose, serum-high (hyperglycemia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sodium, serum-high (hypernatremia) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute graft versus host disease (GVHD) (COH) (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Graft versus host disease (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Veno-Occlusive Disease (VOD) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnea (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation associated with GVHD for BMT studies, if specified in the protocol. (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen I (N=62) | Regimen II (N=17) | Regimen III (N=130) | Regimen IV (N=4) | Regimen V (N=40) | Regimen VI (N=2)
Bone marrow cellularity (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulation - Other (Specify, __) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrinogen (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematemesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin for leukemia studies or bone marrow infiltrative/myelophthisic processes (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/Bleeding - Other (Specify, __) (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Melena/GI bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Prothrombin Time (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion: Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conduction abnormality/atrioventricular heart block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 3 (3) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (3) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Vasovagal episode (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes/flushes (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular surface disease (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision-photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 10 (10) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Diarrhea associated with GVHD for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 3 (3) | 0 (0) | 12 (12) | 0 (0) | 2 (2) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mucositis due to radiation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 0 (0) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 6 (6) | 0 (0) | 15 (15) | 0 (0) | 3 (3) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4) | 0 (0) | 15 (15) | 0 (0) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Insomnia (General disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 5 (9) | 0 (0) | 11 (19) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, __) (General disorders) | 6 (11) | 0 (0) | 10 (18) | 0 (0) | 1 (1) | 0 (0)
Rigors/chills (General disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Sweating (diaphoresis) (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Weight gain - Veno-Occlusive Disease (VOD) for BMT studies if specified in the protocol. (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bilirubin associated with GVHD for BMT studies, if specified in the protocol. (Hepatobiliary disorders) | 3 (3) | 0 (0) | 9 (9) | 0 (0) | 1 (1) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Infections and infestations) | 6 (6) | 0 (0) | 9 (9) | 0 (0) | 3 (3) | 0 (0)
Infection with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L) (Infections and infestations) | 3 (3) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (Specify, __) (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC (Infections and infestations) | 4 (4) | 0 (0) | 8 (8) | 0 (0) | 1 (1) | 0 (0)
Infection without neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Infection, Bacterial (COH) (Infections and infestations) | 3 (5) | 0 (0) | 14 (20) | 0 (0) | 2 (2) | 0 (0)
Infection, Fungal (COH) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection, Viral (COH) (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5 (5) | 2 (2) | 12 (12) | 0 (0) | 2 (2) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 4 (4) | 0 (0) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Acidosis (metabolic or respiratory) (Investigations) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 3 (3) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase (Investigations) | 3 (3) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Alkalosis (metabolic or respiratory) (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Bicarbonate, serum-low (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-high (hypercalcemia) (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calcium, serum-low (hypocalcemia) (Investigations) | 3 (3) | 0 (0) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Investigations) | 2 (2) | 1 (1) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Glucose, serum-high (hyperglycemia) (Investigations) | 6 (6) | 1 (1) | 12 (12) | 0 (0) | 5 (5) | 0 (0)
Glucose, serum-low (hypoglycemia) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Investigations) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Investigations) | 3 (3) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other (Specify, __) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Investigations) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Potassium, serum-high (hyperkalemia) (Investigations) | 2 (2) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Investigations) | 4 (4) | 1 (1) | 10 (10) | 0 (0) | 4 (4) | 0 (0)
Sodium, serum-high (hypernatremia) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sodium, serum-low (hyponatremia) (Investigations) | 3 (3) | 0 (0) | 11 (11) | 0 (0) | 0 (0) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Acute graft versus host disease (GVHD) (COH) (Investigations) | 4 (5) | 0 (0) | 19 (26) | 0 (0) | 2 (3) | 0 (0)
Failure to engraft (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease (Investigations) | 3 (3) | 0 (0) | 17 (18) | 0 (0) | 2 (2) | 0 (0)
Veno-Occlusive Disease (VOD) (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Apnea (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ataxia (incoordination) (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 1 (1) | 8 (8) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Nervous system disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Mood alteration (Nervous system disorders) | 3 (4) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Neurology - Other (Specify, __) (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasms (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (COH) (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sexual/Reproductive Function - Other (Specify, __) (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 11 (11) | 0 (0) | 1 (1) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 8 (8) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 2 (2) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (12) | 0 (0) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation associated with GVHD for BMT studies, if specified in the protocol. (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT00544115/Prot_SAP_000.pdf